CLINICAL TRIAL: NCT00550004
Title: Randomized, Double Blind, Placebo Controlled, Phase 2 Study Evaluating the Efficacy & Safety of RP101 or Placebo in Combination With Gemcitabine Administered as First-Line Treatment to Subjects With Unresectable, Locally Advanced, or Metastatic Pancreatic Adenocarcinoma
Brief Title: Phase II Study to Evaluate Efficacy and Safety of RP101 in Combination With Gemcitabine
Acronym: RP101
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: SciClone Pharmaceuticals (Industry)
Responsible Party: Israel Rios, M.D, Sciclone Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: SCI-RP-Pan-P2-001
Record Dates: First submitted 2007-10-25; First posted 2007-10-26 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2009-10

CONDITIONS: Pancreatic Cancer
Keywords: Unresectable; locally advanced; metastatic pancreatic adenocarcinoma; Stage III; Stage IV
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): RP101 and Gemcitabine
  Interventions: Drug: RP101; Drug: Gemcitabine (1000 mg/m2)
- Arm 2 (Placebo Comparator): Placebo and Gemcitabine
  Interventions: Drug: Gemcitabine (1000 mg/m2)

INTERVENTIONS:
Drug: RP101 — 190 mg oral tablet
  Arms: Arm 1
Drug: Gemcitabine (1000 mg/m2) — 30 minute intravenous infusion
  Other Names: Gemzar

SUMMARY:
This will be a Phase II, multicenter, randomized, double blind, placebo controlled, study of six 28-day treatment cycles for patients with locally advanced, unresectable, or metastatic pancreatic cancer. The study will be conducted at approximately 55 sites in the North American, Europe, and South America. Approximately 153 subjects will be enrolled in a randomization (ratio 2:1).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older
* Not previously treated with chemotherapy for Pancreatic Cancer
* ECOG performance status of 0 or 1
* Life expectancy > 3 months
* Documentation of all sites of pancreatic disease within 28 days prior to randomization
* Adequate hematological, renal, and hepatic function
* Not pregnant or nursing
* Fertile subjects must practice a medically approved method of contraception

Exclusion Criteria:

* Prior history of other malignant tumors
* Participation in another investigational study within 4 weeks prior to treatment start
* Major surgery within 14 days prior to treatment start
* Radiation treatment within 28 days prior to treatment start
* Uncontrolled cardiac atrial or ventricular arrhythmias
* Gastrointestinal tract disease such resulting in an inability to take oral medication
* Known to be seropositive for HIV, HBV, or HCV
* Uncontrolled cancer pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 18 months

SECONDARY OUTCOMES:
Progression Free Survival | 14 months
Evaluate the CA 19-9 levels | 12 months
Compare changes in ECOG | 12 months
Evaluate Safety of RP101 | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Hidalgo, MD, PhD, Study Chair — Centro Integral de Oncologia
Locations (55):
- United States (16):
  - University of Arizona Medical Center, Arizona Cancer Center, Tucson, Arizona
  - Tower Research Foundation at Tower Oncology, Beverly Hills, California
  - University of California at San Francisco, San Francisco, California
  - Integrated Community Oncology Network, LLC, Jacksonville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Gabrail Cancer Center, Canton, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - St. Luke's Cancer Center, Bethlehem, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - South Texas Oncology and Hematology, PA, San Antonio, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Medical College of Wisconsin, Froedtert Multi-Disciplinary Cancer Center, Milwaukee, Wisconsin
- Argentina (3):
  - Hospital Italiano Regional del Sur, Bahía Blanca, Buenos Aires
  - Hospital Británico de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital Zonal General de Agudos San Roque, La Plata, Buenos Aires
- Brazil (5):
  - Hospital de Caridade de Ijuí, Ijuí
  - Hospital de Clínicas de Porto Alegre, Serviço de Oncologia, Porto Alegre
  - Instituto Nacional do Câncer, Rio de Janeiro
  - Núcleo de Oncologia da Bahia, Salvador
  - Hospital do Câncer-AC Camargo, São Paulo
- Chile (2):
  - Fundación Arturo López Pérez, Santiago
  - Hospital Militar, Santiago
- France (3):
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier Départemental, La Roche-sur-Yon
  - Centre Eugene Marquis, Service d'Oncologie Medicale, Rennes
- Germany (3):
  - Universitätsklinikum Dresden, Med. Klinik I, Dresden
  - Klinikum Region Hannover GmbH, Krankenhause Siloah, Hanover
  - Klinikum rechts der Isar, Technische Universität München, München
- Hungary (4):
  - Petz Aladár Megyei Oktató Kórház Orvostovábbképzo Egyetem Oktató-Továbbképzo Kórháza, Onkoradiológia, Gyor, Budapest
  - Fovárosi Önkormányzat Egyesített Szent István és Szent László Kórház-Rendelointézet, Budapest
  - Fovárosi Önkormányzat Uzsoki utcai Kórháza, Budapest
  - Debreceni Egyetem Orvos és Egészségtudományi Centrum, Onkológiai Tanszék, Debrecen
- Maaslandziekenhuis, Sittard, Netherlands
- Peru (3):
  - Hospital Nacional Guillermo Almenara Irigoyen, La Victoria
  - Hospital Nacional Edgardo Rebagliati Martins, Lima
  - Instituto Oncocenter, San Borja
- Poland (4):
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Wojewódzki, Jelenia Góra
  - I Katedra Chirurgii Ogólnej i Klinika Chirurgii Gastroenterologicznej, Krakow
  - Wojewódzki Szpital Specjalistyczny im Kopernika w Lodzi, Lódz
  - Centrum Medyczne MRUKMED, Rzeszów
- Romania (4):
  - Institutul Clinic Fundeni, Bucharest
  - Institutul Oncologic 'Prof. Dr. A. Trestioreanu', Bucharest
  - Spitalul Clinic de Urgenta Floreasca, Bucharest
  - Spitalul Clinic Universitar de Urgenta, Bucharest
- Spain (5):
  - Hospital Universitario Arnau de Vilanova, Servicio de Oncologia, Lleida
  - Centro Integral Oncológico Clara Campal, Hospital de Madrid Norte-San Chinarro, Madrid
  - Hospital 12 de Octubre, Oncology Service, Hospital Materno Infantil, Madrid
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (2):
  - Leicester Royal Infirmary, University Hospitals of Leicester NHS Trust, Leicester, England
  - Mount Vernon Hospital, Middlesex, England

REFERENCES:
- [Derived] Heinrich JC, Tuukkanen A, Schroeder M, Fahrig T, Fahrig R. RP101 (brivudine) binds to heat shock protein HSP27 (HSPB1) and enhances survival in animals and pancreatic cancer patients. J Cancer Res Clin Oncol. 2011 Sep;137(9):1349-61. doi: 10.1007/s00432-011-1005-1. Epub 2011 Jul 22. PMID 21833720
- See also: SciClone Website — http://www.sciclone.com